CLINICAL TRIAL: NCT06005662
Title: Inpatient Buprenorphine Induction With Psilocybin for Opioid Use Disorder: a Randomized Double-blind Trial
Brief Title: Inpatient Buprenorphine Induction With Psilocybin for Opioid Use Disorder
Acronym: BIPOD-In
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was de-prioritized in favor of the similar BIPOD-Out protocol due to a combination of practical considerations and expense. If there are sufficient funds after concluding BIPOD-Out, this study may resume.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00344281
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Psilocybin; Buprenorphine

STUDY DESIGN:
Intervention Model Description: The proposed study is a double-blind, controlled investigation of the effect of 1 high-dose psilocybin (30 mg) session compared to a very low dose session (1 mg) following standard-of-care buprenorphine induction
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and study team will be masked/blinded to intervention.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High-dose psilocybin + buprenorphine (Experimental): High-dose psilocybin (30 mg) session following standard-of-care buprenorphine induction
  Interventions: Drug: Psilocybin
- Very low-dose psilocybin + buprenorphine (Active Comparator): Very low dose psilocybin session (1 mg) following standard-of-care buprenorphine induction
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — The proposed study is a double-blind, controlled investigation of the effect of 1 high-dose psilocybin (30 mg) session compared to a very low dose session (1 mg) following standard-of-care buprenorphine induction on drug abstinence, quality of life, craving, tobacco use, and treatment retention in healthy participants with an active OUD diagnosis
  Other Names: Buprenorphine

SUMMARY:
This study will examine the effect of a single high dose of psilocybin therapy (30 mg) versus a very low dose (1 mg) as an adjunctive therapy to individuals undergoing standard-of-care buprenorphine treatment for Opioid use disorder (OUD). Effects of adjunctive psilocybin will be determined for longitudinal outcomes of opioid abstinence, compliance with buprenorphine maintenance, quality of life, and mood.

DETAILED DESCRIPTION:
The proposed study is a double-blind, controlled investigation of the effect of 1 high-dose psilocybin (30 mg) session compared to a very low dose session (1 mg) following standard-of-care buprenorphine induction on drug abstinence, quality of life, craving, tobacco use, and treatment retention in healthy participants with an active OUD diagnosis. Use of buprenorphine follow standard of care, and the investigators are investigating the additive power of adjunctive psilocybin to enhance opioid abstinence, treatment adherence, quality of life, and mood.

The study will consist of a brief (6-8 day) inpatient phase for standard buprenorphine induction as well as experimental psilocybin administration, an 8-week outpatient phase involving standard buprenorphine maintenance and experimental follow-up meetings, and long-term follow-up sessions for 4 months after. During the inpatient phase, participants will be inducted onto sublingual (SL) buprenorphine (using a buprenorphine/naloxone combination product) while admitted to the Bayview Clinical Research Unit. During this time, participants will also undergo 2-3 preparatory sessions, and will undergo an experimental drug administration session under supportive conditions, during which the participants will receive either a very low dose (1 mg) or a single high (30mg) oral dose of psilocybin under double-blind conditions. At the end of the inpatient phase, participants will be discharged to complete the 8-week outpatient phase, during which participants will undergo visits at 1, 2, 3, 4, 6, and 8 weeks post-dosing session for monitoring of adverse events, clinical status, treatment adherence, and to receive a weekly supply of buprenorphine. All buprenorphine procedures will be open label and will follow standard-of-care practices.

This trial utilizes a Bayesian sequential methodology, employing a maximum sample size of 90 participants and calculating Bayes factors (starting at 20 participants and assessed after each 10) to assess evidence for the null and experimental hypotheses, enabling potential early stopping for efficacy or futility based on predetermined thresholds (Bayes factor of 6 and 1/6). This will be calculated for the primary outcome of opioid abstinence at 8-weeks

ELIGIBILITY:
Inclusion Criteria:

* Age 21-70 years
* Have given written informed consent
* Meet diagnostic criteria for OUD
* No antidepressant medications for approximately 5 half-lives prior to enrollment
* Not currently taking methadone, buprenorphine or naltrexone
* Urine toxicology positive for an opioid
* Has access to stable housing
* Can read, write, and speak English fluently
* Be judged by study team clinicians to be at low risk for suicidality
* Have limited recent use of classic psychedelics (no use in the past year).
* Expresses a desire for sustained recovery from disordered opioid use.

Exclusion Criteria:

General medical exclusion criteria:

* Women who are pregnant, nursing, or not practicing an effective means of birth control
* Cardiovascular conditions: hypertension with resting blood pressure systolic >139 or diastolic >89, angina, heart rate > 99, a clinically significant electrocardiogram abnormality (e.g., atrial fibrillation), Transient Ischemic Attack or Stroke in the last 6 months, peripheral or pulmonary vascular disease, cardiac valvulopathy
* Epilepsy
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking on a daily basis any medications (including herbal substances and supplements) with a central nervous system effect on serotonin, including serotonin-reuptake inhibitors and monoamine oxidase inhibitors.

  o For individuals who have intermittent or as needed use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
* Currently taking efavirenz, Acetaldehyde dehydrogenase inhibitors such as disulfiram (Antabuse), Alcohol dehydrogenase inhibitors, or medicines such as phenytoin, regorafenib, eltrombopag.
* Currently taking buprenorphine, methadone, or naltrexone.
* Unable or unwilling to discontinue acid-reducing agents or major metabolizing enzyme inhibitors for 5-half lives prior to the experimental dosing session.
* Have a seizure disorder, multiple sclerosis, history of significant head trauma, nervous system tumor, movement disorders or any neurodegenerative condition.
* Morbidly obese (>100 pounds above ideal body weight, or Body Mass Index (BMI) >=40, or BMI >=35 with high blood pressure or diabetes)
* Body weight < 45 kilograms
* Be judged by a study team clinician to be at risk for moderate or severe alcohol or benzodiazepine withdrawal.
* Allergic to buprenorphine or hydromorphone
* For blood samples, the following lab values will be exclusionary: transaminases greater than x2 the upper limit of normal lab reference range, hemoglobin less than 11 g/d, and creatinine clearance < 40 ml/min.

Psychiatric Exclusion Criteria:

* Current or past history of meeting diagnostic criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), Bipolar I or II Disorder or Major Depression with psychotic features.
* Have a first or second degree relative with schizophrenia, psychotic disorder (unless substance induced or due to a medical condition), or bipolar I or II disorder.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2027-04 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Opioid Abstinence | up to 8 weeks
  Non-buprenorphine opioid abstinence as verified by urine toxicology at each visit and Timeline Follow Back (TLFB). These will be combined to assess opioid abstinence for each participant. These will be assessed at the 8-week timepoint for the previous 3-weeks. Missing values will be presumed positive.
  Timeline Follow Back (TLFB) for Opioids: This is a self-report of drug use per day. This procedure asks participants to retrospectively quantitate their use of drugs. Greater numbers indicate more days using a substance, smaller numbers or zeros mean less or no days using a substance
  Urine toxicology: Urine samples will be collected at each study visit and screened broadly for illicit drug use including opioids via an outside medical laboratory. Quantitative buprenorphine levels will also be collected following induction to gauge whether buprenorphine is being taken.
  These measurements will be combined to report the number of participants who were abstinent from opioids.
Treatment Retention | 8 weeks
  Treatment retention at 8 weeks, as indicated by participants making all follow-up visits, indicating they are taking buprenorphine and with urine toxicology positive for buprenorphine.
Number of Days Illicit Opioids Used | 8 weeks
  Number of Days Illicit Opioids Used, as indicated by participant self-report and urine toxicology results
Number of Negative Urine Toxicologies | weekly up to 8 weeks
  Number of Negative Urine Toxicologies, as indicated by results from weekly urine toxicologies collected for eight weeks

SECONDARY OUTCOMES:
Quality of Life as assessed by the World Health Organization Quality of Life-BREF (WHOQOL-BREF) | 8 weeks
  World Health Organization Quality of Life-BREF. The WHOQOL produces a multi-dimensional profile of scores across six domains and 24 sub-domains of quality of life, with higher scores representing a greater reported quality of life.
Depression as assessed by the Beck Depression Inventory II (BDII) | 8 weeks
  The Beck Depression Inventory is a multi-item assessment for depression. Scores of 0-10 are considered within normal range, with higher scores representing worsening reported depression.
Anxiety as assessed by the State-Trait Anxiety Inventory (STAI) | 8 weeks
  The State-Trait Anxiety Inventory is a 40-item assessment of state and trait characteristics, with higher scores (more positive items) representing greater severity of mental states such as apprehension, tension, nervousness, and worry.
Number of Participants Abstinent from Other Drug Substances | 8 weeks
  Abstinence from other substances will be measured by combining TLFB and urine toxicology results to report the number of participants who were abstinent from other drug substances

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Nayak, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No